CLINICAL TRIAL: NCT05894616
Title: Home Monitoring and Molecular Phenotyping of Patients With Post-COVID With Focus on Lung Involvement
Acronym: HemCOV
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Michael Runold (Clinical lead), MD, PhD (Unknown); Kristina Piontkovskaya, MD, PhD (Unknown); Björn Nordlund, RN, PhD (Unknown); Angelica Lindén Hirschberg, MD, PhD (Unknown); Tobias Granberg, MD, PhD (Unknown); Karolinska University Hospital (Other); Swedish Heart Lung Foundation (Other); The Swedish Research Council (Other Government); AsthmaTuner AB (Unknown)
Responsible Party: Principal Investigator, Asa Wheelock, Chair, Respiratory Medicine Unit; PhD in Pharmacology and Toxicology, Karolinska Institutet
Other Study IDs: 2022-03768-01
Record Dates: First submitted 2023-06-07; First posted 2023-06-08 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post acute sequale of COVID-19 (PASC): Verified infection with SARS-CoV-2 during wave 1 and 2 (i.e. wild type or alfa variants), prior to 2021-02-28. Diagnosed with post-COVID.
  Experience of dyspnea (mMRC>3 within past 2 weeks) is a required inclusion criteria, with the addition of one of the following: lung obstruction (FEv1/FVC>70 or Z-score < -1.64), lung restriction (FEV1<80% or FVC < 80%, air-trapping, ground glass- or mosaic attenuation observed by HRCT.
- Healthy control recovered from COVID-19: Verified infection with SARS-CoV-2 during wave 1 and 2 (i.e. wild type or alfa variants), prior to 2021-02-28. Fully recovered within 12 weeks of primary infection. No other diagnoses.

SUMMARY:
Post-acute COVID syndrome (PACS) /post-acute sequale of COVID-19 (PASC) / post-COVID is a novel clinical syndrome with unknown biological mechanisms, and to date no standard-of-care, routines for follow-up, or evidence-based treatments have been established. In this project, we will employ a systems medicine approach to identify pathways and networks of genes, proteins and metabolites that are critical in disease onset and progression, towards the goal of understanding specific mechanisms in the etiology of PASC.

The objective of the project is to perform clinical and molecular characterization and sub-phenotyping of patients with PASC, (a.k.a. PACS, or post-COVID), into mechanistically relevant groups, with focus on sex differences in patients with lung involvement. Molecular pathways involved in disease etiology will be identified by correlating rigorous clinical phenotyping and longitudinal eHealth data (home-monitoring via App, home spirometer etc), with multi-molecular level omics profiling of samples collected from the lung, integrated with our systems medicine framework. Aim I involves longitudinal home-monitoring at baseline to investigate fluctuations in general wellbeing, and causes thereof, in PASC patients with lung involvement compared to healthy controls. In Aim II, a set of omics technologies will be employed to provide in-depth molecular characterization of samples from the lung, exhaled particles (PExA), blood and urine. In depth clinical characterizations including photon-counting CT will be performed. In Aim III, integrative statistical- and network modeling approaches will be utilized to: i) identify molecularly distinct sub-groups of obstructive lung diseases based on multi-molecular level network-integration, and ii) identify individual mediators and molecular pathways related to clinical phenotype including longitudinal home-monitoring data, prognosis, diagnosis, and disease etiology of the identified sub-groups.

DETAILED DESCRIPTION:
The core of the home monitoring study is a mobile Application recently developed by our research group. The App, termed HemCOV, is developed on the MyCap/REDCap platformed that is GDPR approved, and is installed on the research subjects (RS) own mobile phone during Visit 1 (virtual visit). The RS will also be assisted in initiate a wearable activity monitor. The RS is then triggered by the App first to answer a set of questionnaires related to health both prior to COVID infection, and currently. Given frequent fatigue among PASC patients, the RS is given 3 days to complete this first task. Thereafter the RS is triggered by the App to answer a brief set of questions daily for 1 weeks to establish a baseline of wellbeing. The RS is then called to Visit 2 which entails spirometry, as well as initiation of a 2 week evaluation using AsthmaTuner (AT). AT triggers the RS to perform spirometry with a portable home spirometer daily. The HemCOV and AsthmaTuner Apps are run daily in parallel for a week. The HemCOV App is the reduced to once every 3 days during the rest of the study to avoid cognitive overload. Initiated and developed by B. Nordlund research group at the Karolinska Institute and Astrid Lindgren Children's Hospital, with support from Swedish innovation programs, AsthmaTuner facilitate asthma diagnosis 7. Given that a number of PASC patients report having been diagnosed with asthma after their initial COVID diagnosis without having been properly investigated, this particular aspect of the AsthmaTuner system is of great interest. In addition, it allows us to follow and identify any alterations in lung function associated with reported alterations in wellbeing, energy levels, or worsening of any PASC-associated symptoms such as fatigue, brain fog, shortness of breath etc. The spirometry registers forced expiratory volume in 1 s (FEV1) and FEV6 (an approximation of forced vital capacity [FVC], to enable the calculation of the ratio that is the basis for measuring lung obstruction (FEV1 / FVC). Visit 3 includes a physical exam by physician to assure the RS is fit to undergo bronchoscopy. If CT has not yet been performed, the RS will also undergo a chest X-ray at this point. In week 4, non-invasive sampling of PExA, blood and urine is performed during Visit 4, and finally in Visit 5 two days later the RS will undergo bronchoscopy, which includes sampling of bronchial epithelial cells (BEC), and immune cells and airway exudates through bronchoalveolar lavage (BAL). Blood hormone profiles to allow investigation of hormone related gender differences in PASC are also performed (lead by endocrinologist prof. Angelica Lindén Hirschberg). Finally at Visit 6, the diffusion capacity is determined. All sample workup and storage of biospecimens will be performed in-house under direct supervision of the PI, utilizing standardized operating procedures (SOP) identical to those utilized in our previous studies, where sample integrity and quality has been confirmed for all omics platforms. Following completion of the base study, participants will be invited for follow-ups after 1, 2, 5 and 10 years. The followup visits include the App questions and questionnaires included in the base study, as well as sampling of blood, urine and PExA.

ELIGIBILITY:
Inclusion Criteria:

PASC group (n=50): Verified SARS-CoV-2 infections (PCR or serology prior to vaccination) during wave 1 and 2 (prior to 2021-02-28). Symptoms >12 weeks after initial illness but with mild-to-moderate disease that did not require hospitalization during the initial infection, disabling persistent symptoms that at some point has affect work capacity 50%. Focus in this study will be placed on subject with some level of lung involvement, including but not limited to Air-trapping on HRCT images, ground glass alterations in radiology, airway obstruction, or shortness of breath as defined by CAT. Experience of dyspnea (mMRC>3 within past 2 weeks) is a required inclusion criteria, with the addition of one of the following: lung obstruction (FEv1/FVC>70 or Z-score < -1.64), lung restriction (FEV1<80% or FVC < 80%, air-trapping, ground glass- or mosaic attenuation observed by HRCT.

Health control group (n=50): Confirmed SARS-CoV-2 infection during wave 1 or 2. Fully recovered within 12 weeks of primary infection.

Exclusion Criteria:

Chronic disease other than asthma. Asthma diagnosis after 2020 allowed in the PASC group.

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Sex at birth
Study Population: See inclusion and exclusion criteria above.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Home monitoring of health status using the eHealth tool HemCOV | 5 weeks
  Home monitoring of symptoms, perceived activity level and actual activity level
Asthma evaluation using AsthmaTuner | 2 weeks
  Spirometry, reversibility test in clinic, followed by FEV1, PEF and variability evaluation using home spirometry
Molecular characterization of particles in exhaled air (PExA) | 2 years
  Collection of PExA material and evaluation of miRNA and proteomes in PEx material
Molecular characterization of samples from the lung collected through bronchoscopy | 2 years
  Analysis of mRNA, miRNA, proteomes, metabolomes, oxylipins and microbiomes from several anatomical locations in the lung

CONTACTS AND LOCATIONS:
Overall Officials: Asa M. Wheelock, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet/Karolinska University Hospital Solna, Stockholm, Sverige, Sweden

IPD SHARING:
Plan to Share IPD: No